CLINICAL TRIAL: NCT02560168
Title: Multidimensional Wavelet Analysis of Surface Electrocardiogram for Identifying Subclinical Myocardial Dysfunction in Patients at Risk for Coronary Artery Disease
Brief Title: Analysis of Surface EKG Signals to Identify Myocardial Dysfunction in Patients at Risk for Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Heart Test Laboratories, Inc. (Industry)
Responsible Party: Principal Investigator, Partho Sengupta, Associate Professor of Medicine and Director of Cardiac Ultrasound Research and Core Lab, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GCO 15-0726; Heart Test Laboratories, Inc. (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; iECG; MyoVista; Heart Test Labs; Wavelet analysis; Surface electrocardiogram
MeSH Terms: conditions — Coronary Artery Disease | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Coronary artery disease (Experimental): Patients scheduled for computed tomographic coronary angiography (CTA)
  Interventions: Device: MyoVista device; Device: Computed tomographic coronary angiography; Device: Transthoracic Echocardiography

INTERVENTIONS:
Device: MyoVista device — MyoVista device is a standard EKG device with additional capabilities in detecting cellular level myocardial electrophysiological signals. The device involves placing leads on the chest, similar to a traditional EKG device
  Other Names: iECG
Device: Computed tomographic coronary angiography — Traditional method of detecting coronary artery disease. CTA will be performed using 64-detector row or higher scanners with electrocardiographic gating in accordance with the Society of Cardiovascular Computed Tomography (SCCT) guidelines. Approximately 80 to 100 ml of intravenous contrast, followed by 50 to 80 ml of saline, will be administered at a rate of 5 ml/s via a power injector through an antecubital vein (on forearm near the elbow).
  Other Names: CTA
Device: Transthoracic Echocardiography
  Other Names: Echocardiogram

SUMMARY:
1. The MyoVista device is capable of detecting surface electrocardiogram signals and sensitive in detecting coronary artery disease compared to traditional computed tomography angiography (CTA)
2. Electrophysiological signals at the cellular level of myocardium are related to specific patterns on the MyoVista device
3. Changes in MyoVista device output and can indicative of future CAD outcomes and need for revascularization

DETAILED DESCRIPTION:
Background Myocardial ischemia is caused by myocardial oxygen supply and demand mismatch. Despite that coronary artery disease (CAD) is the major cause of myocardial ischemia, the symptoms may occur even in the absence of significant CAD. One of the mechanisms suggested for myocardial ischemia in these patients is microvascular ischemia (i.e. mismatch in microscopic vessels), affecting the myocardium (i.e. heart muscle) at the cellular level.

A novel electrocardiographic recording method, the iECG is capable of capturing and amplifying signals from the cellular level that are much lower biologic signals than those processed by a traditional electrocardiogram (ECG). These recordings focus on early detection of myocardial abnormalities by non-linear analysis of electrical activity and physiological phenomenon. This novel assessment might be capable of detecting subclinical myocardial dysfunction in a variety of heart diseases.

Specific Aims

Aim#1: Study the feasibility of detection of CAD using iECG compared to computed tomographic coronary angiography (CTA).

Aim#2: Study the association between patterns of iECG and myocardial dysfunction in patients without CAD compared to echocardiography.

Aim#3: Study the effect of changes in iECG output on future outcomes of CAD and need for revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Sinus rhythms
* Age>18 years
* Both genders

Exclusion Criteria:

* Acute coronary syndromes(ACS)
* Contraindications to the administration of iodinated contrast
* Pregnancy
* Coronary artery bypass surgery (CABG)
* History of cardiac valvular replacement
* Implanted cardiac pacemaker
* Chest deformities
* Unwilling or unable to provide informed consent for study participation
* Enrolled in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Colorized waveform | Day 1
  Spectrum analysis to represent levels and locations of cellular energy and automates the analysis into a simple indication of the level of myocardial abnormality if present.

SECONDARY OUTCOMES:
Change in coronary plaque burden | Baseline and 3 months
  Change in coronary plaque burden at 3 months compared to baseline. Coronary plaque burden will be assessed by assigning a score (0 to 5) according to the SCCT guidelines (0, Normal: absence of plaque and no luminal stenosis; 1, Minimal: plaque with <25% stenosis; 2, Mild: 25% to 49% stenosis; 3, Moderate: 50%to 69% stenosis; 4, Severe: 70% to 99% stenosis; 5, Complete occlusion)
Myocardial wall motion score index (WMSI) | Baseline
  Myocardial wall motion score index (WMSI) will be obtained by dividing the left ventricle into 16 segments7. Each of the segments will be assigned a score that is based on myocardial thickening (1 for Normal or hyperkinetic, 2 for hypokinetic, 3 for akinetic, 4 for dyskinesis, 5 for aneurysmal dilatation). WMSI will be calculated as the sum of scores divided by the number of segments visualized.
Serum electrolytes | 3 months
  Serum electrolytes level to include sodium, potassium, calcium, and magnesium
Serum creatinin level | 3 months
Serum Brain natriuretic peptide (BNP) level | 3 months
Serum cardiac enzymes | 3 months
  Serum cardiac enzymes include creatinin kinase MB fraction (CK-MB)
Serum high sensitivity C-reactive protein (hsCRP) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Partho P Sengupta, MD, DM, FACC, FASE, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States